CLINICAL TRIAL: NCT05015296
Title: A Multicenter, Prospective, Non-interventional Real-world Study of the Impact of Immune Cell Changes During the Perioperative Period on the Prognosis of Patients With Colorectal Cancer
Brief Title: The Impact of Immune Cell Changes During the Perioperative Period on the Prognosis of Patients With Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhongtao Zhang, Director of general surgery, principal investigato, Beijing Friendship Hospital
Other Study IDs: BFH-RWS-CRC
Record Dates: First submitted 2021-07-27; First posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; Immune Cells
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multi-center, prospective, non-interventional real-world study. In a real-world environment, in line with the current status of the domestic diagnosis and treatment process, and on the premise of not increasing the burden of patients and medical resources, we explore the best indicators for predicting the outcome of patients with Clinical Research Coordinator (CRC) after surgery. The inclusion criteria for patients are perioperative patients with CRC. Real-world data analysis were conducted to determine whether immunization interventions versus non-interventions were able to improve patients' clinical outcomes (OS, PFS).

ELIGIBILITY:
Inclusion Criteria:

1. 18-85 years old, regardless of gender;
2. Patients with newly diagnosed CRC who are planned to undergo surgery (including patients with metastases but still feasible for surgery);
3. Patients who have not been diagnosed for the first time and have not received surgical treatment and now planned to undergo surgery(e.g., patients after neoadjuvant radiotherapy and chemotherapy for middle and low rectal cancer).

Exclusion Criteria:

1. Patients who refused to sign informed consent;
2. Patients complicated with other tumors;
3. Pregnant or lactating women;
4. People with a history of psychotropic drug abuse and unable to quit or those with mental disorders;
5. Postoperative histopathological examinations for patients with non-CRC type;
6. Patients who could not be followed up.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. 18-85 years old, regardless of gender;
  2. Patients with newly diagnosed CRC who are planned to undergo surgery (including patients with metastases but still feasible for surgery);
  3. Patients who have not been diagnosed for the first time and have not received surgical treatment and now planned to undergo surgery(e.g., patients after neoadjuvant radiotherapy and chemotherapy for middle and low rectal cancer).
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Changes of immune cells in patients before and after surgery | Postoperative 7 days, 30±7 days, 90 ±10 days, 365 ±30 days
  Preoperative lymphocyte count, postoperative lymphocyte count and normal time, recovery time.
1-year overall survival after surgery | Postoperative 1 year
  the percentage of patients who survived in all patients evaluated at 1 year after surgery
1-year disease-free survival after surgery | Postoperative 1 year
  the percentage of patients who survived disease-free in all patients evaluated at 1 year after surgery
1-year recurrence-free survival after surgery | Postoperative 1 year
  the percentage of patients who survived without recurrence in all patients evaluated at 1 year after surgery